CLINICAL TRIAL: NCT03163563
Title: Perioperative Hypothermia Hypothermia in Ambulatory Surgery by Self-warming or Forced-air Warming Blanket, a Randomised Controlled Trial
Brief Title: Perioperative Hypothermia Hypothermia in Ambulatory Surgery
Status: Completed | Type: Observational
Sponsor: Aleris Helse (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/1481
Record Dates: First submitted 2016-03-02; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Easywarm: Self warming blanket to prevent perioperative hypothermia
  Interventions: Device: Easywarm
- BairHugger: Forced-air warming blanket to prevent perioperative hypothermia
  Interventions: Device: BairHugger

INTERVENTIONS:
Device: Easywarm — Warming blanket
  Groups: Easywarm
Device: BairHugger — Patient warming mattress with continuous warm air.
  Groups: BairHugger

SUMMARY:
The purpose of the study is to measure patient- temperature in the perioperative period of patients undergoing plastic surgery in an ambulatory surgical unit. This study will evaluate if active warming with self-warming blanket (Easywarm®) is as effective as active warming with forced-air blanket (BairHugger®). Second the study will evaluate if one or both methods is effective in preventing perioperative hypothermia.

DETAILED DESCRIPTION:
Background:

Anesthesia medicaments given in general anesthesia cause impaired thermoregulation and thermogenesis. After induction of general anesthesia the core temperature is reduced to redistribution of blood from the body core to the cooler skin. Later impaired thermogenesis contributes to further loss of heat.

Mild hypothermia (<36 degrees Celsius) contributes to increased incidence of wound infections, prolonged stay in the post anesthesia care unit, shivering and reduced patient comfort.

There are several effective interventions to prevent hypothermia such as active warming pre-, per- and postoperatively. Preheated intravenous fluids and medical interventions to alter the blood distribution from the periphery to the body core have been effective in preventing hypothermia.

In the department both self-warming blanket (Easywarm®) and forced-air blanket (BairHugger®) are routinely used to prevent hypothermia. It has been observed that a few patients undergoing plastic surgery with anesthesia time more than one hour are shivering and feeling cold in the postoperative period.

Purpose:

The purpose of the study is to observe and measure patient- temperature in the perioperative period of patients undergoing plastic surgery in an ambulatory surgical unit. This study will evaluate if active warming with self-warming blanket (Easywarm®) is as effective as active warming with forced-air blanket (BairHugger®). Second the study will evaluate if one or both methods is effective in preventing perioperative hypothermia.

Design:

The is a quality assurance study deigned as a prospective randomised trial. With a validated non-invasive termometer (SpotOn® 3M) temperature is measured before, during and after surgical procedures in general anesthesia. An equal number of notes with the number 1 and 2 were put into an envelope (1=EasyWarm®, 2=BairHugger®). For each operation theater a note is drawn, and all patients in that operation theater receives active warming according to the number on the note.

Population data:

Sex, age , weight, height, BMI, medication, morbidities and ASA class will be registered.

Measurements:

* temperature (Celsius)
* Blood pressure
* Heartrate
* SaO2
* Temperature-comfort "numeric rating scale" (NRS)

Other registrations:

* Medicines given during the study period.
* Start and end of anesthesia and surgery
* Time when temperature is above or eual to 36 degrees Celsius.
* Time when the patient go home

Data is collected and registered on a dataform. Data are analysed in a anonymized excel workbook.

ELIGIBILITY:
Inclusion Criteria:

* Patients for planned plastic surgery with duration of general anesthesia ≥ 60 minutes.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for plastic surgery with planned total anestesia for more than 60 minutes are enrolled consecutively.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Temperature | Perioperative period
  Temperature Celsius measured by SpotOn 3M

SECONDARY OUTCOMES:
Medication given during study period | Perioperative period
  Type and dosage is registered. Ephedrine and phenylephrine are known to interact with temperature regulation.
Temperature Numerical Rating Scale | Perioperative period.
  To identify at which temperature the patient is comfortably warm without need for warming intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stig S Tyvold, MD PhD, Principal Investigator — Aleris Helse AS
Locations (1):
- Aleris Solsiden, Trondheim, Sør-Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tyvold SS. Preventing hypothermia in outpatient plastic surgery by self-warming or forced-air-warming blanket: A randomised controlled trial. Eur J Anaesthesiol. 2019 Nov;36(11):843-850. doi: 10.1097/EJA.0000000000001087. PMID 31567576